CLINICAL TRIAL: NCT06539481
Title: A Non-randomised, Open-label, Uncontrolled, Multi-centre, Phase IIIb Study Evaluating the Safety and Efficacy of Fluocinolone Acetonide 190 Micrograms Intravitreal Implant in Paediatric Subjects From 6 Years to Less Than 18 Years With Recurrent Non-infectious Uveitis Affecting the Posterior Segment of the Eye
Brief Title: Open Label Trial Studying the Safety and Effectiveness of ILUVIEN® (190μg) in Children and Adolescents, Who Have Recurrent Non-infectious Uveitis Affecting the Posterior Segment of the Eye.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alimera Sciences (Industry)
Responsible Party: Sponsor
Organization: ANI Pharmaceuticals (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ALI-P01-21-006
Record Dates: First submitted 2024-07-30; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Non-infectious Uveitis Affecting the Posterior Segment of the Eye

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ILUVIEN® 190μg (Experimental)
  Interventions: Drug: fluocinolone acetonide 190 micrograms

INTERVENTIONS:
Drug: fluocinolone acetonide 190 micrograms — ILUVIEN®, is a tiny tube that is to be implanted in the eye and releases low levels of the corticosteroid (fluocinolone acetonide) in the eye. ILUVIEN® delivers corticosteroid directly to the intended site of action for up to 36 months.

SUMMARY:
The main aim is to test how safe and effective the medicine ILUVIEN® (190μg) is for children and adolescents, who have non-infectious uveitis that keeps coming back and affects the back of the eye.

The main thing Alimera wants to find out is how well the implant works for treating non-infectious uveitis in the back of the eye. Treatment success will be measured after 6 months of using the implant.

The treatment will be considered successful if two things happen:

1. No swelling in the back of the eye called cystoid macular oedema;
2. A decrease in the cloudiness inside the eye, called vitreous haze, by at least two levels compared to how it was before the treatment, or the vitreous haze is completely gone.

Participants will:

1. Receive a single treatment with ILUVIEN®, which is a tiny tube that is to be implanted in the eye and releases low levels of the corticosteroid (fluocinolone acetonide) in the eye for up to 36 months.
2. Be followed for 36 months for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* Males and females of ≥6 and <18 years of age at time of consent
* Non-infectious posterior, intermediate or panuveitis in the study eye with a history of recurrence ≥1 per year as assessed by the Investigator
* Uveitis in the study eye not adequately controlled by the preferred standard of care due to intolerable adverse effects or poor response, in the judgment of the Investigator
* Treatment with systemic corticosteroid or other systemic therapies given for at least 3 months within the previous 12 months prior to Day 1

Exclusion Criteria:

* History of intraocular surgery in the study eye within 90 days of the screening visit.
* Hypersensitivity to FA or any component of ILUVIEN®
* History of any form of glaucoma or ocular hypertension in study eye, unless study eye has been previously treated with an incisional IOP-lowering surgical procedure at least 90 days prior to the screening visit and that procedure has resulted in stable IOP in the normal range (10-21 mmHg)
* Increased intraocular pressure >25 mmHg or that required treatment including increases in medications, surgery (other than drainage surgery), or hospitalisations, within 4 weeks prior to baseline that, in the opinion of the Investigator, would pose an unacceptable risk to the patient participating in the study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2024-08-31 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Absence of cystoid macular oedema on Optical Coherence Tomography and a decrease from baseline in vitreous haze grade of ≥2 steps, or absence of vitreous haze. | 6 months after administration
  The primary endpoint for evaluating the effect of the implant on non-infectious uveitis affecting the posterior segment of the eye will be based on treatment success, determined at 6 months after administration. Treatment success will be determined based on a composite variable defined as Absence of cystoid macular oedema on Optical Coherence Tomography and a decrease from baseline in vitreous haze grade of ≥2 steps, or absence of vitreous haze.
Rate of cataract formation and Rate of IOP elevation | 6 months after administration
  The primary endpoint for evaluating the safety of the implant on non-infectious uveitis affecting the posterior segment of the eye will be determined.
  * Rate of cataract formation
  * Rate of IOP elevation (Change from baseline in IOP and incidence of significant changes in IOP, including: IOP>21 mmHg, IOP>25 mmHg, IOP>30 mmHg, increases from baseline of 10 mmHg or more).

SECONDARY OUTCOMES:
Changes in vision and incidence of increase in IOP, AE, and uveitis recurrence | Every 6 months over 3 years
  * Absence of CMO and decrease from baseline in vitreous haze grade of ≥2 steps, or absence of vitreous haze at end of the study
  * Uveitis recurrence rate following treatment, compared to the uveitis recurrence rate over the 12 months prior to enrolment
  * Incidence of recurrence of non-infectious uveitis affecting the posterior segment in the SE and in the FE after receiving study treatment
  * Time to recurrence of non-infectious uveitis affecting the posterior segment
  * Change in macular oedema,
  * Change in BCVA
  * Change in vitreous haze
  * Change in AC cell grade
  * Incidence of secondary increase in IOP and secondary increase in IOP requiring surgical intervention
  * Incidence and onset of secondary lens opacity and extraction
  * Number of adjunctive treatments required to treat recurrences of uveitis
  * Presence of active chorioretinal
  * Presence of retinal vascular lesions
  * Incidence of ocular infection
  * Incidence of AEs
  * Change from baseline in cup-to-disc ratio
Incidence of secondary increase in IOP, secondary increase in IOP requiring surgical intervention, and ocular and non-ocular AEs. | 3, 6, 12, and 36 months.
  Mandatory safety measures including IOP checks will be performed every 3 months.
  The following secondary safety endpoints will be assessed at 6 months, 12 months or 36 months
  * Incidence of secondary increase in IOP
  * Incidence of secondary increase in IOP requiring surgical intervention
  * Incidence of ocular and non-ocular AEs.

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (2):
  - Charité - Universitätsmedizin Berlin Institute of Health Department of Ophthalmology, Berlin
  - Augenzentrum am St. Franziskus-Hospital Münster, Münster
- Spain (2):
  - Hospital Universitario Cruces, Bilbao
  - Fundación Jiménez Díaz, Madrid
- United Kingdom (2):
  - University of Bristol Bristol Medical School, Bristol
  - Sheffield Teaching Hospitals NHS Foundation Trust and Sheffield Children NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No